CLINICAL TRIAL: NCT01163864
Title: Affect Regulation Training for Pregnant Smokers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Clara Bradizza, Senior Research Scientist, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Q607; R01DA021802 (NIH)
Record Dates: First submitted 2010-07-13; First posted 2010-07-16 (Estimated); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Smoking Cessation
Keywords: smoking; smoking relapse; smoking cessation; pregnancy; smoking cessation in pregnant women
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- affect regulation training (Experimental)
  Interventions: Behavioral: affect regulation training
- health and lifestyle (Active Comparator)
  Interventions: Behavioral: health and lifestyle

INTERVENTIONS:
Behavioral: affect regulation training — 8 sessions of a 1-hour long treatment intended to help women deal more effectively with negative affect; cognitive-behavioral smoking cessation intervention
  Arms: affect regulation training
Behavioral: health and lifestyle — 8 sessions of a 1-hour long treatment designed to help women improve their overall health; cognitive-behavioral smoking cessation intervention
  Arms: health and lifestyle

SUMMARY:
Recent data indicate that approximately one-third of women of childbearing age smoke cigarettes, and 25-50% of women smoke during pregnancy. Cigarette smoking during pregnancy is a significant public health issue that can have profound effects on women's health and the health of their developing fetus. Smoking among pregnant women is associated with high levels of negative affect, which play a key role in the maintenance of smoking behavior and in difficulty quitting smoking during pregnancy. Despite the clear role of negative affect in the maintenance of smoking among pregnant women, and while this issue has received increased attention by clinicians and researchers, the investigators know of no smoking cessation intervention that combines coping skills and emotion regulation approaches to address the role of negative affect in smoking cessation. Smoking cessation treatment strategies that have demonstrated effectiveness in regular smokers have not translated into effective treatment strategies for pregnant women, particularly low-income pregnant women. The goal of this project is to develop and test an affect regulation smoking cessation intervention for low-income pregnant smokers.

The major aims of this project will be addressed in two sequential phases. In Phase 1, the investigators will develop two 8-session smoking cessation treatment manuals including: (a) Affect Regulation Training plus Cognitive-Behavioral Treatment (ART+CBT) and (b) a Health and Lifestyle plus Cognitive-Behavioral Treatment (HLS+CBT) control intervention. In Phase 2, the investigators will conduct a randomized clinical trial pilot study (Total N = 60) to compare the ART+CBT and HLS+CBT conditions on: a) the feasibility and acceptability of the interventions, (b) the impact of these interventions (ART+CBT and HLS+CBT) on smoking cessation rates at the end of the 8 treatment sessions (these occur approximately 2 months after treatment initiation) and at the 6-month post-quit date assessment (Session 2 is the quit date), (c) affect regulation skills, and (d) negative affect among pregnant smokers. The long-term goal of this proposed research is to increase smoking cessation rates among pregnant smokers, which would provide significant long-term health benefits for both mothers and their infants. This Stage 1 application will be used to generate feasibility and preliminary efficacy data, setting the stage for a Stage II efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age,
* pregnancy involving single birth,
* less than 24 weeks pregnant,
* negative affect smoker,
* smoking at least 1 cigarette per day,
* no substance abuse diagnosis except marijuana,
* no more than .50 ounces of ethanol per day,
* can provide a collateral to verify smoking information.

Exclusion Criteria:

* acute psychosis,
* lack of familiarity with the English language.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2007-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
smoking cessation rate using the Timeline Followback Interview for smoking | end of 8 session treatment (about 2 months after treatment initiation)
  We will compare the number of women who are abstinent from smoking in the ART+CBT group vs. the HLS+CBT group using the Timeline Followback Interview for smoking

SECONDARY OUTCOMES:
smoking cessation rate using the Timelineline Followback Interview for smoking | 6-month post-quit date (Session 2 is always the quit date)
  We will compare the number of women who are abstinent from cigarettes in the ART+CBT group vs. the HLS+CBT group using the Timeline Followback Interview for smoking
treatment feasibility | end of 8-session treatment
  We will compare the number of women who complete the 8-session treatment in the ART+CBT vs. he HLS+CBT group.
treatment acceptability | end of 8-session treatment
  We will compare the treatment ratings by participants for the ART+CBT group vs. the HLS+CBT group using the Treatment Acceptability Questionnaire
affect regulation skills | end of 8-session treatment
  We will compare the scores on measures of affect regulation skills of ART+CBT group vs. HLS+CBT group using the Difficulties in Emotion Regulation Scale (DERS).
negative affect | end of 8-session treatment
  We will compare levels of negative at the end of treatment of the ART+CBT group vs. the HLS+CBT group using both Positive and Negative Affect Scale

CONTACTS AND LOCATIONS:
Overall Officials: Clara Bradizza, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- Research Institute on Addictions, University at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Derived] Fillo J, Kamper-DeMarco KE, Brown WC, Stasiewicz PR, Bradizza CM. Emotion regulation difficulties and social control correlates of smoking among pregnant women trying to quit. Addict Behav. 2019 Feb;89:104-112. doi: 10.1016/j.addbeh.2018.09.033. Epub 2018 Sep 26. PMID 30286396
- See also: Research Institute on Addiction website — http://www.ria.buffalo.edu/
- See also: Description of project on institutional website — http://www.ria.buffalo.edu/currproj.html